CLINICAL TRIAL: NCT04953130
Title: Adding Male Single Dose HPV Vaccination to Female HPV Vaccination in Tanzania
Acronym: Add-Vacc
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Mwanza Intervention Trials Unit, National Institute for Medical Research (Unknown); York Biomedical Research Institute, Hull York Medical School, University of York (Unknown); Cancer Epidemiology Research Programme Institut Català d' Oncologia (Unknown); Karolinska Institute Department of Laboratory Medicine (Unknown); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MITU-003
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: HPV Infection; Vaccine Preventable Disease
MeSH Terms: conditions — Papillomavirus Infections; Vaccine-Preventable Diseases

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial with 26 communities (13 per arm)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Male vaccination + national HPV vaccination programme (Experimental): Single dose of the 4-valent HPV vaccine (Gardasil®; Merck & Co.) offered to all eligible boys aged 14 to 18 years in the 13 intervention communities. Girls aged 14 years are offered 2 doses of Gardasil® through the Tanzanian national HPV vaccine programme
  Interventions: Biological: Gardasil® HPV vaccine
- National HPV vaccination programme only (Active Comparator): Girls aged 14 years are offered 2 doses of Gardasil® through the Tanzanian national HPV vaccine programme
  Interventions: Biological: Gardasil® HPV vaccine

INTERVENTIONS:
Biological: Gardasil® HPV vaccine — Single dose 4-valent HPV vaccine in males. Gardasil®, manufactured by MSD, consists of a licensed prophylactic virus-like particle (VLP) vaccine that protects against 4 HPV genotypes (HPV 6, 11, 16, 18).
  Other Names: 4-valent HPV vaccine

SUMMARY:
Add-Vacc is an unblinded cluster-randomised trial (CRT) with two arms: (i) the national HPV vaccination programme (girls aged ~14 years, control arm) and (ii) the national programme plus single-dose male HPV vaccination given to a multi-year cohort of boys (intervention arm). The CRT will be conducted in 26 communities/clusters (13 per arm) in northern Tanzania. Boys aged 14 to 18 years in the intervention arm will receive one dose of the 4-valent HPV vaccine (Gardasil®) that protects against HPV 6, 11, 16, and 18. Population genital HPV prevalence in 18 to 21-year-olds will be compared between intervention clusters (female and male vaccination) and control clusters (female vaccination only) at 3 years after the intervention. Blood sampling for immune responses and adverse event data collection will be performed in a subset of 200 male subjects in selected intervention clusters.

ELIGIBILITY:
Inclusion Criteria:

* Parents and adult male participants (aged 18 years) must sign an ICF and male participants aged less than 18 years must sign an informed assent form (IAF), indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study and to receive HPV vaccination. If the parent or participant cannot read or write, the procedures must be explained and informed consent/assent must be witnessed by a literate third party who is not involved in the conduct of the study.
* Participants must have been born male, and must be aged 14 to 18 years inclusive at time of vaccination.
* Participants must be living in an intervention community (cluster).
* Participants must be willing and able to comply with the protocol requirements.
* Participants must agree to avoid all non-trial immunisations in the 14 days following vaccination with the trial vaccine, other than emergency vaccinations such as post-exposure rabies or tetanus vaccinations.
* Participants must be healthy as determined by a medical history. A physical examination will be conducted if necessary according to the clinician's judgement.

Exclusion Criteria:

Boys will be excluded from HPV vaccination if:

* They have previously been vaccinated against HPV.
* They have a history of allergy or anaphylaxis to one or more of the HPV vaccine components, to yeast or to latex.
* They are enrolled in another vaccine research study that specifically specifies that they must not participate in a study of another vaccine
* They have been diagnosed with a chronic condition (except HIV, as per the comment above), such as an autoimmune condition, sickle cell disease, degenerative disease, neurologic or genetic disease, among others;
* There are significant conditions or clinically significant findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., it would compromise their safety or well-being).

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10400 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Impact of adding single-dose male HPV vaccination to the national HPV vaccination programme in girls on population 4-valent HPV genotype prevalence in 18 to 21-year-old females and males | Month 36
  Prevalence of 4-valent vaccine HPV genotype DNA (HPV 6, 11, 16 or 18) in males and females aged 18 to 21 years in intervention clusters and control clusters 36 months post-male vaccination

SECONDARY OUTCOMES:
Immunogenicity and safety of single dose 4-valent HPV vaccination in boys | Month 12, 24 and 36
  Proportion seroconverting to, and geometric mean antibody titres (GMTs) for, HPV vaccine genotypes, and safety and tolerability (local and systemic adverse events), measured in a subset of 200 vaccinated boys
Impact of female-only vaccination through the national vaccination programme on population HPV prevalence in 18 to 21-year-old males and females | Month 36
  The proportion of females, and of males, aged 18 to 21 years in the control arm with detectable genital 4-valent HPV vaccine genotype DNA at baseline and at M36.
Uptake of dose 1 and coverage of dose 2 in eligible target groups for the national HPV vaccination programme; | Month 36
  The proportion of females aged 16 years who received 1 dose of HPV vaccine (uptake) and who complete 2 doses (coverage) by arm at baseline and M36
Acceptability of a gender-neutral approach to HPV vaccination | Month 24
  Self-reported acceptability of and barriers to receiving male vaccination by community members and to delivering male HPV vaccination by health care workers (HCW)
Cost-effectiveness of adding a multi-year single dose male HPV vaccination strategy to the national female HPV vaccination programme | Month 36
  Incremental cost-effectiveness ratio for single dose male vaccination plus existing female vaccination programme compared to female vaccination only

CONTACTS AND LOCATIONS:
Locations (1):
- Mwanza Intervention Trials Unit, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263